CLINICAL TRIAL: NCT00640016
Title: A Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Efficacy, Safety, and Tolerability of CAT-354
Brief Title: A Study to Assess the Efficacy, Safety, and Tolerability of CAT-354 in Subjects With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prematurely by the sponsor due to slow recruitment.
Sponsor: MedImmune LLC (Industry)
Collaborators: Cambridge Antibody Technology (Other); PRA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAT-354-0603; 2007-002090-31 (EudraCT Number)
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Asthma
Keywords: Asthma; CAT-354; Tralokinumab
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo matched to CAT-354 intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Interventions: Other: Placebo
- CAT-354 1 mg/kg (Experimental): CAT-354 1 milligram per kilogram (mg/kg) of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Interventions: Biological: CAT-354 1 mg/kg
- CAT-354 5 mg/kg (Experimental): CAT-354 5 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Interventions: Biological: CAT-354 5 mg/kg
- CAT-354 10 mg/kg (Experimental): CAT-354 5 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56
  Interventions: Other: CAT-354 10 mg/kg

INTERVENTIONS:
Other: Placebo — Placebo matched to CAT-354 intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: Placebo
Biological: CAT-354 1 mg/kg — CAT-354 1 milligram/kilogram (mg/kg) of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: CAT-354 1 mg/kg
Biological: CAT-354 5 mg/kg — CAT-354 5 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Other Names: Tralokinumab
  Arms: CAT-354 5 mg/kg
Other: CAT-354 10 mg/kg — CAT-354 10 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
  Arms: CAT-354 10 mg/kg

SUMMARY:
To investigate the effects of CAT-354 on airway hyper-responsiveness (AHR) in uncontrolled asthma.

DETAILED DESCRIPTION:
This is a randomized, stratified, double-blind, placebo-controlled, multicenter, multinational study in subjects with uncontrolled asthma despite optimal treatment. Following confirmation of eligibility, subjects will be randomly assigned on Day 0, to 1 of 4 dose groups 1 mg/kg CAT-354, 5 mg/kg CAT-354, 10 mg/kg CAT or Placebo to match all doses of CAT-354. Doses of the assigned treatment will be administered on three occasions 28 days apart. Subjects will be assessed for efficacy, including airway hyper-responsiveness (AHR), safety, pharmacokinetic, pharmacodynamics and immunogenicity until Day 84 post-first dose.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent is obtained prior to any study related procedure taking place
* Women either infertile (example [e.g.], hysterectomized, sterile or post-menopausal with amenorrhea of least 1 year duration) or who are practicing an acceptable form of birth control
* Uncontrolled (refractory) asthma despite treatment with a minimum dose of 800 microgram (mcg) beclomethasonedipropionate or equivalent inhaled corticosteroid per day plus 1 or more additional controller, that is, long-acting beta-agonist, leukotriene antagonist or theophylline. Oral corticosteroids (not parenteral) as additional treatment at any dose are acceptable
* A forced expiratory volume in 1 second (FEV1) acceptable for airway hyper-responsiveness (AHR) challenge tests (greater than 60 percent of predicted normal) on the challenge days
* A provocative concentration of methacholine causing a 20 percent fall in FEV1 (PC20) less than 4 milligram per milliliter (mg/mL)
* Aged 18-80 years
* A 12-lead electrocardiogram (ECG) with no-clinically significant abnormalities
* Clinical chemistry, hematology and urinalysis results within the laboratory reference ranges or deemed not clinically significant by the Investigator
* Body weight of less than 130 kilogram (kg)
* No other clinically significant abnormality on history and clinical examination
* Able to comply with the requirements of the protocol.

Exclusion Criteria:

* Experienced a severe exacerbation within 28 days preceding Day -28/-14 to Day 0
* Onset of uncontrolled seasonal allergy symptoms within 28 days preceding Day -28/-14 to Day 0
* Subjects with a history of allergic rhinitis, seasonal allergy or esophagitis must be optimally controlled and remain on a stable treatment regimen during the study
* Participation in another study within 5 half-lives or 3 months of the start of this study, whichever is the longer
* Lower respiratory tract infection within 6 weeks of Day -28/-14 to Day 0
* Current smokers or ex-smokers with greater than 10 pack-years
* Blood donation (more than 550 mL) in the previous 2 months
* Excessive intake of alcohol (as judged by the Investigator) or evidence of drug or solvent abuse
* Subjects with a physician-diagnosis of any other significant lung disease, including a primary diagnosis of chronic obstructive pulmonary disease or bronchiectasis, or lung cancer, sarcoidosis, tuberculosis, pulmonary fibrosis and cystic fibrosis
* Concurrent medication from Day -28/-14 to Day 0 (Screening visit) and for the duration of the study with any of the prohibited medications
* Significant, uncontrolled disease including serious psychological disorders, chronic renal failure, uncontrolled hypertension
* systolic blood pressure greater than 200 millimeters of mercury (mmHg), or diastolic blood pressure greater than 100 mmHg, heart disease, psoriasis requiring treatment and subjects who have had a heart attack or stroke within the 3 months preceding Day -28/-14 to Day 0, or who have a known aneurysm
* Onset of uncontrolled seasonal allergy symptoms within 28 days preceding Day -28/-14 to Day 0
* Subjects with a history of allergic rhinitis, seasonal allergy or esophagitis must be optimally controlled and remain on a stable treatment regimen during the study
* Any factor which, in the opinion of the Investigator, would jeopardize the evaluation or safety or be associated with poor adherence to the protocol (that is, inability to complete study diary, perform peak expiratory flow (PEF) measurements)
* The subject's primary care physician recommends the subject should not take part in the study
* Known hypersensitivity to CAT-354 or its components, to the challenge agents used in the study or to related drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Mayer, M.D., Study Director — PRA Health Sciences
Locations (41):
- Australia (9):
  - St. Vincents Hospital, Thoracic Medicine Unit, Darlinghurst, New South Wales
  - Respiratory Medicine Department, Mater Adult Hospital,, South Brisbane, Queensland
  - Princess Alexandria Hospital, Dept of Respiratory Medicine, Woolloongabba, Queensland
  - Eastern Clinical Research Unit, Box Hill, Victoria
  - Monash Medical Centre, Dept Respiratory Medicine., Clayton, Victoria
  - Dep of Respiratory & Sleep Medicine, Western Hospital, Footscray, Victoria
  - Respiratory & Sleep Medicine, Royal Melbourne Hospital, Parkville, Victoria
  - Lung Institute WA, Sir Charles Gardner Hospital, Nedlands, Western Australia
  - WA Lung Research, Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Germany (11):
  - Evangelische Lungenklinik Berlin - Kardiologie/Pneumologie - 1.OG, Haus 23, Berlin
  - Med. Klinik m. S. Infektiologie und Pneumologie, Charite - Universitätsmedizin Berlin, Berlin
  - Lungen und Bronchialheikunde, Bonn
  - Praxis für Lungen-und Bronchialheilkunde, Allergologie und Umweltmedizin, Bonn
  - Rheinische Friedrich-Wilhelms-Universität, Medizinische Klinik und Poliklinik II, Innere Medizin, Bonn
  - Internistisches Facharztzentrum Stresemannallee, Frankfurt
  - Universitätsklinikum Magdeburg Fachbereich Pneumologie, Magdeburg
  - Universitätsklinikum Mainz, Klinische Forschung Pneumologie, III. med. Klinik, Mainz
  - Universitätsklinikum Münster Klinik und Poliklinik für Dermatologie, Münster
  - Universität Rostock, Medizinische Fakultät Klinik und Poliklinik für Innere Medizin, Rostock
  - Johanniter-Krankenhaus im Fläming gGmbH, Pneumologie, Treuenbrietzen
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Poland (10):
  - ISPL Centrum Medyczne, Bialystok
  - Prywatny Gabinet Internistyczno-Alergologiczny, Bialystok
  - Samodzielny Publiczny Centralny Szpital Kliniczny Slaskiej Akademii Medycznej, Klinika Pneumologii, Katowice
  - Niepubliczny Zakład Opieki Zdrowotnej Atopia, Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 Im. Norberta Barlickiego w Łodzi, Lodz
  - Szpital ZOZ Lubin Oddzial Alergologiczny i Chorob Wewnetrznych, Lubin
  - Wojewodzki Szpital Specjalistyczny, Poradnia Alergologiczna, Lublin
  - Alergopneuma Przychodnia Alergologiczno-Pulmonologiczna Marek Michnar i wsp., Lublin
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
  - Wojewódzki Szpital Specjalistyczny w Zgierzu, Zgierz
- United Kingdom (10):
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Gartnavel General Hospital, Glasgow
  - University Hospitals of Leicester NHS Trust, Glenfield Hospital, Leicester
  - Royal Brompton Hospital, London
  - University Hospital of South Manchester NHS Foundation Trust, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Gwent Hospital, Newport
  - Norfolk and Norwich University Hospital, Norwich
  - Lister Hospital, Stevenage, Hertfordshire

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Started | 3 | 3 | 4 | 4
Treated | 3 | 2 | 4 | 4
Completed | 1 | 1 | 1 | 1
Not Completed | 2 | 2 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Study termination | 2 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.00 (11.136) | 34.00 (14.933) | 37.75 (9.878) | 40.75 (15.086) | 37.00 (11.708)
Gender [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 3 | 11
  Male | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Doubling Concentration of Methacholine at Day 28
Description: Change in doubling concentrations of methacholine was calculated as Log2 PC20 (Visit x) - Log2 PC20 (Baseline), where x was the post-baseline assessment (Day 28) and PC20 was provocative concentration of methacholine causing 20 percent fall in forced expiratory volume in 1 second (FEV1). FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Change in doubling concentration was summarized for sub-therapeutic dose (placebo and CAT-354 1 milligram/kilogram [mg/kg]) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: Baseline and Day 28
Population: Safety population included all participants who received at least 1 dose of study medication. Here 'n' signifies those participants who were evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: log2 milligram/deciliter (mg/dL)
Groups:
- Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg): CAT-354 5 mg/kg or 10 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
- Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg): Placebo or CAT-354 1 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 8 | 5
log2 milligram/deciliter (mg/dL)
  Baseline (n=8, 5) | -0.604 (2.4080) | -1.545 (0.8952)
  Change at Day 28 (n=5, 4) | -0.207 (1.0450) | 0.125 (2.3433)

2. Secondary Outcome: Change From Baseline in Doubling Concentration of Methacholine at Day 56, 84 or Early Termination
Description: Change in doubling concentrations of methacholine was calculated as Log2 PC20 (Visit x) - Log2 PC20 (Baseline), where x was the post-baseline assessment (Day 28) and PC20 was provocative concentration of methacholine causing 20 percent fall in forced expiratory volume in 1 second (FEV1). FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Change in doubling concentration was summarized for sub-therapeutic dose (placebo and CAT-354 1 mg/kg) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: Baseline, Day 56, 84 or early termination (any time before Day 84)
Population: Safety population included all participants who received at least 1 dose of study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure, and 'n' signifies those participants who were evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: log2 mg/dL
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 3 | 2
log2 mg/dL
  Change at Day 56 (n=2, 2) | 0.062 (1.1309) | -1.423 (0.4059)
  Change at Day 84 (n=2, 2) | -0.038 (0.1410) | -1.846 (0.0431)
  Change at Early termination (n=3, 2) | -0.514 (0.8636) | 0.417 (0.9840)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: The FEV1 was maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FEV1 was summarized for sub-therapeutic dose (placebo and CAT-354 1 mg/kg) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: Predose, 30 minutes and 6 hours post-end of infusion on Day 0, 28 and 56; Day 4, 14, 35, 63, 84 or early termination (any time before Day 84)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 8 | 5
liters
  Day 0: Predose (n=8, 5) | 2.718 (0.5458) | 2.640 (0.3994)
  Day 0: 30 minutes postdose (n=8, 5) | 2.684 (0.5695) | 2.624 (0.4126)
  Day 0: 6 hours postdose (n=8, 5) | 2.606 (0.5731) | 2.550 (0.4304)
  Day 4 (n=8, 5) | 2.814 (0.6048) | 2.606 (0.2919)
  Day 14 (n=6, 5) | 2.323 (0.5703) | 2.520 (0.0812)
  Day 28: Predose (n=5, 4) | 2.598 (0.4676) | 2.850 (0.2082)
  Day 28: 30 minutes postdose (n=4, 4) | 2.535 (0.5639) | 2.918 (0.2822)
  Day 28: 6 hours postdose (n=4, 4) | 2.400 (0.5254) | 2.665 (0.2748)
  Day 35 (n= 4, 4) | 2.260 (0.5464) | 2.778 (0.4228)
  Day 56: Predose (n=2, 2) | 2.555 (0.6718) | 2.700 (0.3677)
  Day 56: 30 minutes postdose (n=2, 2) | 2.705 (0.7990) | 2.830 (0.1697)
  Day 56: 6 hours postdose (n=2, 2) | 2.510 (0.7071) | 2.690 (0.2404)
  Day 63 (n= 2, 2) | 2.505 (0.6859) | 2.580 (0.0283)
  Day 84: (n=2, 2) | 2.680 (0.7778) | 2.540 (0.4101)
  Early Termination (n=4, 3) | 3.018 (0.5803) | 2.867 (0.4400)

4. Secondary Outcome: Forced Vital Capacity (FVC)
Description: The FVC was volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. FVC was summarized for sub-therapeutic dose (placebo and CAT-354 1 mg/kg) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: as for outcome 3
Population: Safety population included all participants who received at least 1 dose of study medication. Here, 'n' signifies those participants who were evaluable for this measure at specified time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 8 | 5
liters
  Day 0: Predose (n= 8, 5) | 3.828 (0.8215) | 3.666 (0.6068)
  Day 0: 30 minutes postdose (n= 8, 5) | 3.823 (0.6500) | 3.722 (0.6752)
  Day 0: 6 hours postdose (n= 8, 5) | 3.808 (0.7718) | 3.722 (0.7297)
  Day 4 (n= 8, 5) | 3.988 (0.6058) | 3.824 (0.7415)
  Day 14 (n=6, 5) | 3.462 (0.5926) | 3.710 (0.5220)
  Day 28: Predose (n=5, 4) | 3.908 (0.7670) | 3.883 (0.6412)
  Day 28: 30 minutes postdose (n=4, 4) | 3.878 (0.7876) | 3.980 (0.7951)
  Day 28: 6 hours postdose (n=4, 4) | 3.810 (0.7409) | 3.790 (0.4830)
  Day 35 (n=4, 4) | 3.613 (0.6874) | 3.920 (0.7777)
  Day 56: Predose (n=2, 2) | 3.700 (0.5233) | 3.410 (0.3818)
  Day 56: 30 minutes postdose (n=2, 2) | 3.775 (0.5303) | 3.540 (0.4667)
  Day 56: 6 hours postdose (n=2, 2) | 3.715 (0.6435) | 3.545 (0.3748)
  Day 63 (n=2, 2) | 3.705 (0.5162) | 3.575 (0.5020)
  Day 84: (n=2, 2) | 3.710 (0.6505) | 3.415 (0.3323)
  Early Termination (n=4, 3) | 3.908 (0.8070) | 4.193 (0.8364)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) as Percentage of Forced Vital Capacity (FVC)
Description: Percentage of FEV1 was calculated as (FEV1/FVC)*100. It signified the percentage of the total amount of air exhaled from the lungs during the first second of forced exhalation. FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. Result was summarized for sub-therapeutic dose (placebo and CAT-354 1 mg/kg) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: Predose, 30 minutes and 6 hours post-end of infusion on Day 0, 28 and 56; Day 4, 14, 35, Day 63, 84 or early termination (any time before Day 84)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of FVC
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 8 | 5
percentage of FVC
  Day 0: Predose (n=8, 5) | 71.875 (10.3156) | 72.600 (11.4149)
  Day 0: 30 minutes postdose (n=8, 5) | 70.250 (9.1613) | 71.600 (13.1833)
  Day 0: 6 hours postdose (n=8, 5) | 69.125 (12.5178) | 69.600 (12.1984)
  Day 4 (n=8, 5) | 71.000 (13.1909) | 69.400 (8.7063)
  Day 14 (n=6, 5) | 66.667 (7.5011) | 68.800 (8.1670)
  Day 28: Predose (n=5, 4) | 67.400 (13.1263) | 74.500 (11.2694)
  Day 28: 30 minutes postdose (n=4, 4) | 66.500 (13.9881) | 74.500 (9.6782)
  Day 28: 6 hours postdose (n=4, 4) | 63.750 (12.3390) | 71.250 (13.8173)
  Day 35 (n=4, 4) | 62.500 (7.5498) | 71.750 (7.8049)
  Day 56: Predose (n=2, 2) | 68.000 (8.4853) | 80.000 (19.7990)
  Day 56: 30 minutes postdose (n=2, 2) | 71.000 (11.3137) | 81.000 (15.5563)
  Day 56: 6 hours postdose (n=2, 2) | 67.000 (7.0711) | 76.500 (14.8492)
  Day 63 (n=2, 2) | 66.500 (9.1924) | 72.500 (9.1924)
  Day 84 (n=2, 2) | 71.500 (9.1924) | 75.500 (19.0919)
  Early Termination (n=4, 3) | 77.750 (9.8107) | 69.000 (5.5678)

6. Secondary Outcome: Asthma Control Questionnaire (ACQ) Total Score
Description: The ACQ is questionnaire that comprises of 7-questions evaluating participant's asthma control. Six self-administered questions assess asthma control over the past week covering nocturnal waking, morning symptoms, activity limitations, shortness of breath, wheezing, and short-acting bronchodilator use; using 7-point ordinal rating scale from 0 (good control) to 6 (poor control). Seventh question is completed by a health professional on forced expiratory volume in 1 second (FEV1) percentage (%) predicted; scale: 0 (greater than [>] 95% predicted) to 6 (less than [<] 50% predicted. Final score is the average score of the 7 questions, with a score range of 0 (well controlled) to 6 (extremely poor controlled). Result was summarized for sub-therapeutic dose (placebo and CAT-354 1 mg/kg) and therapeutic dose (CAT-354 5 mg/kg and CAT-354 10 mg/kg), as per planned analysis.
Time Frame: Baseline, Day 28, 56, 84 or early termination (any time before Day 84)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 8 | 5
units on a scale
  Baseline (n=8, 5) | 2.44 (0.737) | 1.77 (0.861)
  Day 28 (n=5, 4) | 2.00 (0.416) | 1.46 (0.914)
  Day 56 (n=2, 2) | 1.43 (0.808) | 1.50 (1.111)
  Day 84 (n=2, 2) | 1.57 (1.010) | 2.36 (0.101)
  Early Termination (n=5, 3) | 1.72 (1.304) | 0.57 (0.378)

7. Secondary Outcome: Post-bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: The FEV1 was maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.
Time Frame: Day 0 to 84
Population: Data was not collected and hence, not analyzed for this outcome measure because the study was prematurely terminated on the basis of several factors namely, observed low rate of participant randomisation into the study; delay caused by temporary halt of study and potential for expiry date of investigation medicinal product before end of study.
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Diary Data
Description: Participants recorded asthma symptoms, use of reliever inhalers (beta-agonist use for symptom relief and as prophylaxis), and morning and evening peak expiratory flow (PEF) measurements in a diary.
Time Frame: Day 0, 4, 14, 28, 35, 56, 63 to Day and 84
Population: as for outcome 7
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Exacerbations
Description: Exacerbation was defined as: Mild (determined from diary data) - 2 consecutive days satisfying the same or 1 of the following criteria: any night with awakening(s) due to asthma or morning PEF 20 % or more below baseline where baseline = average of the 10 days before randomization or as-needed medication use of 2 inhalations or more in 24 hours above baseline where baseline = average of the 10 days before randomization. Severe (determined by taking an exacerbation update and history): deterioration of asthma resulting in emergency treatment or hospitalization or need for oral steroids for 3 days or more (as judged by the Investigator).
Time Frame: Day 0 to Day 84
Population: as for outcome 7
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Morning Peak Flow and Peak Flow Variability
Description: Peak flow is a participant's maximum speed of expiration.
Time Frame: Day 0 to Day 84
Population: as for outcome 7
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Adult Asthma Quality of Life (QoL) Questionnaire Final Score
Description: The AQLQ: a 32-item questionnaire evaluating quality of life of participants with asthma including 4 domains (symptoms, activity limitations, emotional function, and environmental stimuli). Participants are asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean response to all questions. The 4 domain scores are the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment).
Time Frame: Day 0, 28, 84 or early termination (any time before Day 84)
Population: as for outcome 7
Arm/Group | Therapeutic-dose (CAT-354 5mg/kg and CAT-354 10mg/kg) | Sub-therapeutic Dose (Placebo or CAT-354 1mg/kg)
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for CAT-354
Time Frame: Predose, 10 minutes and 6 hours post-end of infusion on Day 0, 28 and 56
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study medication and had sufficient post-dose blood samples to estimate Cmax. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
microgram/milliliter (mcg/mL)
  After first dose (Day 0) | 27.7 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 219 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 163 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After second dose (Day 28) | 34.5 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 255 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 235 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After third dose (Day 56) | 33.4 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 338 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 251 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

13. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) for CAT-354
Time Frame: Predose, 10 minutes and 6 hours post-end of infusion on Day 0, 28 and 56
Population: PK population included all participants who received at least 1 dose of study medication and had sufficient post-dose blood samples to estimate Cmax. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
mcg/mL
  After first dose (Day 0) | 4.84 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 51.8 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 52.8 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After second dose (Day 28) | 7.91 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 54.1 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 64.4 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After third dose (Day 56) | 9.70 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 85.5 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 68.4 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

14. Secondary Outcome: Area Under the Serum Concentration Time Curve From Time Zero to Last Measurable Concentration (AUC [0 - t]) for CAT-354
Time Frame: Predose, 10 minutes and 6 hours post-end of infusion on Day 0, 28 and 56
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: microgram*day/milliliter (mcg*day/mL)
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
microgram*day/milliliter (mcg*day/mL)
  After first dose (Day 0) | 335 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 2820 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 2090 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After second dose (Day 28) | 408 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 4720 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3080 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  After third dose (Day 56) | 499 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3690 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 3420 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

15. Secondary Outcome: Accumulation Ratio for CAT-354 (RA)
Description: Accumulation ratio (RA) is calculated for Cmax, Cmin and AUC as RA for Cmax = Cmax (56 - 84)/Cmax (0 - 28); Similarily, RA for Cmin = Cmin (56 - 84)/Cmin (0 - 28) and RA for AUC= AUC (56 - 84)/AUC (0 - 28) where Cmax (0 - 28) and Cmax (56 - 84) are the maximum observed serum concentration after first dose (Day 0 to Day 28) and after third dose (Day 56 to Day 84), respectively; Cmin (0 - 28) and Cmin (56 - 84) are the minimum observed serum concentration after first and third dose, respectively; AUC (0 - 28) and AUC (56 - 84) are the area under the serum concentration time curve over a dosage interval determined after first and third dose, respectively.
Time Frame: Predose, 10 minutes and 6 hours post-end of infusion on Day 0, 28 and 56
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- CAT-354 1 mg/kg: CAT-354 1 mg/kg of body weight intravenous infusion over 60 minutes on Day 0, 28 and 56.
Arm/Group | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 1 | 1 | 1
ratio
  RA for Cmin | 1.20 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.54 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.73 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  RA for Cmax | 2.00 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.65 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.30 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.
  RA for AUC | 1.49 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.31 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group. | 1.64 (NA) — Standard deviation was not estimable because only 1 participant was evaluable in this reporting group.

16. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 84 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 0 to 84
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Number analyzed (Participants) | 3 | 2 | 4 | 4
participants
  TEAEs | 2 | 2 | 4 | 3
  TESAEs | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Day 0 to 84
Arm/Group | Placebo | CAT-354 1 mg/kg | CAT-354 5 mg/kg | CAT-354 10 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 2/3 | 2/2 | 4/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | CAT-354 1 mg/kg (N=2) | CAT-354 5 mg/kg (N=4) | CAT-354 10 mg/kg (N=4)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | CAT-354 1 mg/kg (N=2) | CAT-354 5 mg/kg (N=4) | CAT-354 10 mg/kg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Forced expiratory volume decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was prematurely terminated due to low recruitment rate, delay due to temporary halt and potential for expiry date of study drug. It was not considered possible to draw meaningful conclusions from the small dataset.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The Principal Investigator (PIs) also agree for data to be presented first as a joint, multi-center publication.